CLINICAL TRIAL: NCT02707653
Title: Sublingual Misoprostol for the Treatment of Incomplete Abortion: Operations Research
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Department of Medical Research, Lower Myanmar (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001
Record Dates: First submitted 2016-02-19; First posted 2016-03-14 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Incomplete Abortion
MeSH Terms: conditions — Abortion, Incomplete | interventions — Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Miso (Other): Misoprostol 400 s/l
  Interventions: Drug: Misoprostol

INTERVENTIONS:
Drug: Misoprostol — 400 mcg sublingual misoprostol
  Other Names: cytotec

SUMMARY:
This study will investigate the use of misoprostol for first-line treatment of incomplete abortion at tertiary hospitals in Myanmar.

DETAILED DESCRIPTION:
This open-label feasibility study seeks to examine the potential of 400μg sublingual misoprostol for the treatment of incomplete abortion provided at tertiary hospitals.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed incomplete abortion
2. No known contraindications to the study drug
3. Uterine size no larger than 12 weeks at time of presentation for care
4. No signs of severe infection, defined as at least two of the following:

   * foul smelling discharge,
   * fever > 38 degrees C, 100 degrees Fahrenheit
   * uterine tenderness.
5. No hemodynamic disturbances (pulse >110/min and systolic bp <100)
6. General good health
7. Agree to comply with study procedures including return for follow up visit
8. Live or work within one hour from a study site
9. Willing and able to sign consent forms

Exclusion Criteria:

1. Inability to provide informed consent

Ages: 12 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 75 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage of women with complete uterine evacuation with study medication alone. | 14 days

SECONDARY OUTCOMES:
Percentage of women experiencing side effects | 7-14 days
  occurrence of side effects, if any, including fever, chills, nausea, vomiting, headache, diarrhea, and pain.
Level of self-reported acceptability of treatment | 7-14 days
  Woman's satisfaction with the treatment, woman's likelihood to use the treatment in the future, woman's likelihood of recommending the treatment to a friend, providers' satisfaction with the treatment, likelihood provider would recommend the treatment in a similar situation.

CONTACTS AND LOCATIONS:
Locations (2):
- Burma (2):
  - Central Woman's Hospital, Yangon
  - Thingyan Sanpya Hospital, Yangon

IPD SHARING:
Plan to Share IPD: Undecided